CLINICAL TRIAL: NCT04531657
Title: Influenza Vaccine Antibody Response and 6-month Persistence in Lung Transplant Recipients Using Two Definitions of Seroprotection
Brief Title: Influenza Vaccine in Lung Transplant Patients - Seroprotection
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0240e; A561000 (Other: UW Madison); PHARM/PHARMACY/PHARMACY (Other: UW Madison); 2009-0002 (Registry Identifier: Institutional Review Board)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Influenza
Keywords: Post-lung transplant; Healthy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccine, Post-transplant: Cohort consist of individuals who have received lung transplants Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- Vaccine, Healthy Control: Cohort consists of healthy individuals who received the influenza vaccine Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine

INTERVENTIONS:
Drug: Influenza vaccine — influenza vaccine 0.5 ml intramuscularly during 2008-2009 season for measurement of A/Brisbane/59/2007(H1N1)-like, A/Brisbane/10/2007(H3N2)-like, and B/Florida/4/2006-like antigens

SUMMARY:
This a sub-study of a 5-year study designed to investigate how antibody and T cell responses following influenza vaccine compare among lung transplant patients, patients waiting for lung transplantation, and healthy individuals.

This study is designed to investigate two different definitions of influenza vaccine seroprotection at mid-season in lung transplant patients.

DETAILED DESCRIPTION:
Given the significant risk of morbidity and mortality, it is critical and highly recommended that lung transplant patients receive annual influenza immunizations that confer protection throughout the influenza season. Previous studies have demonstrated that transplant recipients and nonimmunocompromised populations display similar rates of seroprotection between 3 and 5 weeks after influenza vaccination, despite the transplant population achieving generally lower antibody concentrations. Two studies show influenza vaccine antibody persistence at reasonable rates at 1 year, but not 2 years, after immunization. However, there are no studies comparing seroprotection rates 6 months after vaccination, reflecting adequate coverage throughout the entire influenza season.

Seroprotection has traditionally been defined as an antibody concentration of at least 40 hemagglutination units (HAU) after vaccination, which is the criterion for influenza vaccine licensure. This concentration of antibody provides protection from infection at a rate of about 50% in typically healthy individuals. Protection from infection improves with higher antibody concentrations. For this study, a HAU of at least 160 was selected as a more conservative definition of seroprotection, where protection may reach up to 95%.

The hypothesis is that seroprotection, defined as 40 HAU or greater, will persist up to 6 months at high rates in lung transplant patients and that these rates will be comparable to the rates in healthy individuals. As a secondary outcome, seroprotection rates are compared when 160 HAU or greater was used to define seroprotection.

Influenza vaccine responses in lung transplant patients and healthy control subjects without lung disease will be compared over the course of the 2008 to 2009 influenza season.

Serum collected from participants before immunization, 2 to 4 weeks after immunization (postimmunization), and 6 months after immunization.

[This substudy that was originally registered to NCT00205270 and subsequently registered to its own NCT number for the purpose of clarity in linked results]

ELIGIBILITY:
Inclusion Criteria:

* Receiving care post-lung transplant at University of Wisconsin Hospital
* Healthy adult

Exclusion Criteria:

* Allergy to eggs
* Moderate to severe febrile illness
* Active treatment for acute rejection
* Received season's influenza vaccine prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult or patient receiving care post-lung transplant at University of Wisconsin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Seroprotection to Influenza Vaccine: 40 HAU | up to 6 months
  The hypothesis is that seroprotection, defined as 40 HAU or greater, will persist up to 6 months at high rates in lung transplant patients and that these rates will be comparable to the rates in healthy individuals. Seroprotection (antibody titer greater than or equal to 1:40) will be reported for H1N1, H3N2, and B viral antigens.

SECONDARY OUTCOMES:
Number of Participants with Seroprotection to Influenza Vaccine: 160 HAU | up to 6 months
  Seroprotection (antibody titer greater than or equal to 1:160) will be reported for H1N1, H3N2, and B viral antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Long AJ, Worzella SL, Moran JJ, Hayney MS. Influenza vaccine antibody response and 6-month persistence in lung transplant recipients using two definitions of seroprotection. Transplantation. 2015 Apr;99(4):885-9. doi: 10.1097/TP.0000000000000391. PMID 25148380